CLINICAL TRIAL: NCT04786691
Title: How do You Take Your Coffee Before Anesthesia: A Randomized Controlled Crossover Study Comparing Gastric Emptying With Black Coffee vs Coffee With Cream
Brief Title: How do You Take Your Coffee Before Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 262000
Record Dates: First submitted 2021-03-03; First posted 2021-03-08 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia; Aspiration; Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Crossover
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators performing the gastric ultrasound will be blinded to which arm of the study the participant is currently in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Black coffee first (Placebo Comparator): 12 oz of black coffee with no additives is the first intervention tested
  Interventions: Other: Addition of half and half to coffee; Other: Addition of non-dairy creamer to coffee; Other: Black
- Coffee with half and half first (Active Comparator): 12 oz of black coffee with 1 oz of half and half is the first intervention tested
  Interventions: Other: Addition of half and half to coffee; Other: Addition of non-dairy creamer to coffee; Other: Black
- Coffee with non-dairy creamer first (Active Comparator): 12 oz of black coffee with 1 oz of liquid non-dairy creamer is the first intervention tested
  Interventions: Other: Addition of half and half to coffee; Other: Addition of non-dairy creamer to coffee; Other: Black

INTERVENTIONS:
Other: Addition of half and half to coffee — 1 oz of half and half is added to 12 oz of black coffee and given to participants assigned to this arm after the baseline gastric ultrasound
Other: Addition of non-dairy creamer to coffee — 1 oz of non-dairy creamer is added to 12 oz of black coffee and given to participants assigned to this arm after the baseline gastric ultrasound
Other: Black — No Creamer

SUMMARY:
Undergoing anesthesia requires patients to fast pre-operatively to allow the stomach to empty and prevent aspiration pneumonia but patients are allowed to drink "clear" liquids up to 2 hours before surgery. Clear liquids are defined as water, carbonated sodas, black coffee or tea without milk or sugar, and juices without pulp. Many Americans prefer to take their coffee with half and half or coffee creamer rather than black. This study will determine whether the addition of a small amount of cream to coffee makes any difference to the volume in the stomach after 2 hours.

This study will use healthy volunteers as study participants. Each participant will participate in the study 3 times with at least 2 days in between. We will use a bedside ultrasound machine to measure their stomach content volume at baseline and then they will consume one of 3 different prepare drinks - black coffee, coffee with half and half, or coffee with non-dairy coffee creamer. After 2 hours, we will scan their stomach again and measure stomach content volume and compare it to the first measurement. The participants will repeat this two more times on different days so that they would have had a chance to consume all three prepared coffee drinks in a random order.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65

Exclusion Criteria:

* Diabetes mellitus
* Delayed gastric emptying
* Previous gastric surgery
* Lactose intolerance
* Current pregnancy
* Consumption of solid/liquids in 6 hours prior to commencement of ultrasound study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Yeh, MBBS, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-Black Coffee, 2-half and Half, 3-creamer: 12 oz of black coffee with no additives is given to participants assigned to this arm first after the baseline gastric ultrasound. Based on the randomization order, participants will then participate in the coffee with half and half arm and then the coffee with non-dairy creamer arm.
- 1-Black Coffee, 2-creamer, 3-half and Half: 12 oz of black coffee with no additives is given to participants assigned to this arm first after the baseline gastric ultrasound. Based on the randomization order, participants will then participate in the coffee with non-dairy creamer arm then coffee with half and half.
- 1-half and Half, 2-black Coffee, 3-creamer: 12 oz of black coffee with 1 oz of half and half is given to participants assigned to this arm first after the baseline gastric ultrasound. Based on the randomization order, participants will then participate in the black coffee arm and the coffee with non-dairy creamer arm.
- 1-half and Half, 2-creamer, 3-black Coffee: 12 oz of black coffee with 1 oz of half and half is given to participants assigned to this arm first after the baseline gastric ultrasound. Based on the randomization order, participants will then participate in the coffee with non-dairy creamer arm then the black coffee arm.
- 1-creamer, 2-black Coffee, 3-half and Half: 12 oz of black coffee with 1 oz of liquid non-dairy creamer is given to participants assigned to this arm first after the baseline gastric ultrasound. Based on the randomization order, participants will then participate in the black coffee arm then the coffee with half and half arm.
- 1-creamer, 2-half and Half, 3-black Coffee: 12 oz of black coffee with 1 oz of liquid non-dairy creamer is given to participants assigned to this arm first after the baseline gastric ultrasound. Based on the randomization order, participants will then participate in the coffee with half and half arm then the black coffee arm.
Period: First Intervention (2 Hours)
Arm/Group | 1-Black Coffee, 2-half and Half, 3-creamer | 1-Black Coffee, 2-creamer, 3-half and Half | 1-half and Half, 2-black Coffee, 3-creamer | 1-half and Half, 2-creamer, 3-black Coffee | 1-creamer, 2-black Coffee, 3-half and Half | 1-creamer, 2-half and Half, 3-black Coffee
Started | 2 | 3 | 2 | 4 | 3 | 4
Completed | 2 | 3 | 2 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (2 Days)
Arm/Group | 1-Black Coffee, 2-half and Half, 3-creamer | 1-Black Coffee, 2-creamer, 3-half and Half | 1-half and Half, 2-black Coffee, 3-creamer | 1-half and Half, 2-creamer, 3-black Coffee | 1-creamer, 2-black Coffee, 3-half and Half | 1-creamer, 2-half and Half, 3-black Coffee
Started | 2 | 3 | 2 | 4 | 3 | 4
Completed | 2 | 3 | 2 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (2 Hours)
Arm/Group | 1-Black Coffee, 2-half and Half, 3-creamer | 1-Black Coffee, 2-creamer, 3-half and Half | 1-half and Half, 2-black Coffee, 3-creamer | 1-half and Half, 2-creamer, 3-black Coffee | 1-creamer, 2-black Coffee, 3-half and Half | 1-creamer, 2-half and Half, 3-black Coffee
Started | 2 | 3 | 2 | 4 | 3 | 4
Completed | 2 | 3 | 2 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (2 Days)
Arm/Group | 1-Black Coffee, 2-half and Half, 3-creamer | 1-Black Coffee, 2-creamer, 3-half and Half | 1-half and Half, 2-black Coffee, 3-creamer | 1-half and Half, 2-creamer, 3-black Coffee | 1-creamer, 2-black Coffee, 3-half and Half | 1-creamer, 2-half and Half, 3-black Coffee
Started | 2 | 3 | 2 | 4 | 3 | 4
Completed | 2 | 3 | 2 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (2 Hours)
Arm/Group | 1-Black Coffee, 2-half and Half, 3-creamer | 1-Black Coffee, 2-creamer, 3-half and Half | 1-half and Half, 2-black Coffee, 3-creamer | 1-half and Half, 2-creamer, 3-black Coffee | 1-creamer, 2-black Coffee, 3-half and Half | 1-creamer, 2-half and Half, 3-black Coffee
Started | 2 | 3 | 2 | 4 | 3 | 4
Completed | 2 | 3 | 2 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants were randomized to receive all 3 interventions of consumption of black coffee, coffee with half and half, and coffee with non-dairy creamer.
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18
Body Mass Index [Median (Full Range); unit: kg/m^2] | 22.4 [20.1 to 34.1]

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Gastric Volume Post Coffee Consumption Compared to the Baseline Gastric Volume
Description: Gastric volume calculated based on measured cross-sectional area (CSA) of gastric antrum and participant's age. CSA is measured at baseline after fasting for 6 hours and measured again 2 hours after consuming prepared coffee drink
Time Frame: Baseline 6 hours after fasting and 2 hours after intervention
Measure: Mean (95% Confidence Interval); unit: milliliters
Groups:
- Black Coffee: 12 oz of black coffee with no additives given to participants after the baseline gastric ultrasound either as the first, second, or third intervention.
- Coffee With Half and Half: 12 oz of black coffee with 1 oz of half and half given to participants after the baseline gastric ultrasound either as the first, second, or third intervention.
- Coffee With Non-dairy Creamer: 12 oz of black coffee with 1 oz of liquid non-dairy creamer given to participants after the baseline gastric ultrasound either as the first, second, or third intervention.
Arm/Group | Black Coffee | Coffee With Half and Half | Coffee With Non-dairy Creamer
Number analyzed (Participants) | 18 | 18 | 18
milliliters | 13 [-0.6 to 26.6] | 5 [-8.6 to 18.6] | -1.5 [-15.1 to 12.1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 3 month period
Description: This study was low risk for serious adverse events and all-cause mortality. The collection approach for adverse events was through non-systematic assessment.
Arm/Group | Black Coffee | Coffee With Half and Half | Coffee With Non-dairy Creamer
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT04786691/Prot_SAP_000.pdf